CLINICAL TRIAL: NCT01540643
Title: Zenith® Spiral-Z® AAA Iliac Leg Graft Post-market Registry
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-015
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Abdominal Aortic Aneurysm; Aorto-iliac Aneurysm
Keywords: abdominal aortic aneurysm; iliac leg graft
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Abdominal aortic aneurysm
  Interventions: Device: Iliac Leg Graft

INTERVENTIONS:
Device: Iliac Leg Graft — Zenith® Spiral-Z® AAA Iliac Leg Graft

SUMMARY:
The purpose of this registry is to obtain case reports of physician experience with the Spiral-Z® graft under routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Patient is implanted with Zenith® Spiral-Z® AAA Iliac Leg Graft.

Exclusion Criteria:

* Patients for whom this device would not normally be considered standard of care.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with an FDA approved Zenith® Spiral-Z® AAA Iliac Leg Graft
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assess short term and longer term outcomes, including outcomes related to patency, of the Zenith® Spiral-Z® AAA Iliac Leg Graft. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lindsay, Principal Investigator — Toronto General Hospital
Locations (31):
- United States (27):
  - Valley Vascular Consultants, Huntsville, Alabama
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami Hospital, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University Hospital, Augusta, Georgia
  - Missouri Heart Center, Columbia, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - St. Vincent's Heart and Vascular Center, Billings, Montana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albany Medical Center Hospital, Albany, New York
  - Westchester Medical Center, Hawthorne, New York
  - Mount Sinai Hospital, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Mount Carmel East, Columbus, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - St. Luke's University Hospital, Bethlehem, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Physican's Regional Medical Center, Knoxville, Tennessee
  - Houston VA, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Providence Regional Medical Center Everett, Everett, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Froedert Hospital, Milwaukee, Wisconsin
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Civic Campus, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Lindsay T, Jazaeri O, Sherman SM, Saunders AT, Forbes TL; Spiral-Z Registry Investigators. Final results from a postmarket registry of an iliac leg graft with a continuous, spiral nitinol stent. J Vasc Surg. 2020 Aug;72(2):576-583.e1. doi: 10.1016/j.jvs.2019.10.078. Epub 2020 Jan 19. PMID 31964568